CLINICAL TRIAL: NCT03910153
Title: Effect of MSPrebiotic Digestion Resistant Starch on Gastrointestinal Function and Blood Glucose Levels
Brief Title: Effect of MSPrebiotic on Gastrointestinal Function and Blood Glucose Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MSP Starch Products Inc. (Industry)
Collaborators: Source Nutraceutical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MSPCT2
Record Dates: First submitted 2019-04-05; First posted 2019-04-10 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Gastrointestinal Function
Keywords: Prebiotic; Potato Starch; Resistant Starch; MSPrebiotic; Gut Health; Microbiome; Glucose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo - (Age 30-50 years) (Placebo Comparator)
  Interventions: Other: Placebo
- MSPrebiotic - (Age 30-50 years) (Experimental)
  Interventions: Dietary Supplement: MSPrebiotic
- Placebo - (Aged 70 years and above) (Placebo Comparator)
  Interventions: Other: Placebo
- MSPrebiotic - (Aged 70 years and above) (Experimental)
  Interventions: Dietary Supplement: MSPrebiotic

INTERVENTIONS:
Dietary Supplement: MSPrebiotic — MSPrebiotic digestion resistant starch from potatoes (30 g) will be mixed in 1 glass (approximately 250 mL) of non-heated fluid or non-heated semi solid food and consumed. If the subject is on any medications, the potato resistant starch will be administered either 2 hours before medications or 2 hours after participants have taken their medications.
  Arms: MSPrebiotic - (Age 30-50 years); MSPrebiotic - (Aged 70 years and above)
Other: Placebo — Corn starch (30 g) will be mixed in 1 glass (approximately 250 mL) of non-heated fluid or non-heated semi solid food and consumed. If the subject is on any medications, the corn starch will be administered either 2 hours before medications or 2 hours after participants have taken their medications.
  Arms: Placebo - (Age 30-50 years); Placebo - (Aged 70 years and above)

SUMMARY:
The objective of the study is to investigate the impact of daily consumption of MSPrebiotic at a dosage level of 30 g per day for 12 weeks on gastrointestinal microbiota in the elderly (> 70 years age) and another age group (30 to 50 years). In addition, impact of MSPrebiotic on short chain fatty acids, glucose and insulin levels as well as metabolomic changes will also be studied. A randomized, double-blinded study will be conducted to assess the health benefits of MSPrebiotic and compared with a placebo. This study will provide substantiation for a beneficial effect of MSPrebiotic resistant starch on gut microbiome.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent (or by the authorized 3rd party).
* Willing to provide stool (2 times) and blood (6 times) samples over the 14 week study period
* Subjects between 30-50 and above 70 years of age
* Subjects willing to provide fasting blood during Screening and weeks 0, 2, 6, 10 and 14 visits
* Female subjects not pregnant or breast feeding
* Female subjects not planning for pregnancy during the study period

Exclusion Criteria:

* Crohn's disease or any other inflammatory bowel disease
* Individuals with Lupus, or on cancer chemotherapy
* Pre-diabetes or Diabetes
* Thyroid disease
* Renal disease
* Hepatic disease
* Previous gastrointestinal surgery (intestinal resection, gastric bypass, colorectal surgery)
* Subjects on probiotic (e.g. yoghurt),
* Subjects on antibiotics at time of recruitment or on antibiotics within the previous five weeks
* Individuals experiencing dysphagia
* Subjects using additional fiber supplements
* Subjects on digestants, emetics and antiemetics, medications for acid peptic disease and antacids.
* Subjects allergic to potato or corn
* Have conditions, factors, medication (other than those listed above) that the Investigator believes may affect the response of the gut or the interpretation of the test results

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2019-04-08 (Actual); Primary Completion 2019-10-07 (Actual); Study Completion 2019-10-07 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in gut microbiome | 0 and 14 weeks
  Gut microbiome composition (ratio between number of Firmicutes and Bacteroides) will be measured using 16S ribosomal ribonucleic acid (rRNA) gene sequencing in stool samples
Changes from baseline in concentration of short chain fatty acids in stool samples | 0 and 14 weeks
  Concentration of short chain fatty acids (acetate, propionate, butyrate, isobutyrate, valerate,isovalerate) in feces will be measured using gas chromatographic method
Changes from baseline in bowel movements with respect to number of bowel movements and stool consistency | 0, 2, 6,10 and 14 weeks
  Number of bowel movements will be measured using questionnaire. Stool consistency will be measured using questionnaires recording Bristol score. Bristol stool chart indicates the following types: Type 1-Separate hard lumps, like nuts; Type 2-Sausage-shaped but lumpy; Type 3-Like a sausage but with cracks on its surface; Type 4-Like a sausage or snake, smooth and soft; Type 5-Soft blobs with clear-cut edges (passed easily); Type 6-Fluffy pieces with ragged edges, a mushy stool; Type 7-Watery, no solid pieces. Entirely liquid.
Changes from baseline in blood glucose concentrations | 0, 2, 6,10 and 14 weeks
  Blood glucose levels concentrations will be measured using standard laboratory methods
Changes from baseline in blood insulin concentrations | 0 and 14 weeks
  Blood insulin concentrations will be measured using standard laboratory methods

SECONDARY OUTCOMES:
Changes from baseline in tolerability in terms of excessive flatulence, abdominal pain, and bloating: questionnaires | 0, 2, 6,10 and 14 weeks
  Tolerability of consuming MSPrebiotic in terms of excessive flatulence, abdominal pain, and bloating will be measured using questionnaires. The questionnaire will record the severity of flatulence, abdominal pain and bloating on a scale of 1 to 5 where 1=none and 5=extreme.
Changes from baseline in overall health in terms of outpatient visits and hospitalizations | 0, 2, 6,10 and 14 weeks
  Overall health will be measured using questionnaires on outpatient visits and hospitalizations. The questionnaire contains Yes/No question to record if the subject had any outpatient visits or hospitalizations.
Changes from baseline in concentration of blood lipids and C-reactive protein Inflammatory marker C-reactive protein. Metabolomic changes | 0 and14 weeks
  Concentration of blood lipids and C-reactive protein will be measured using standard laboratory methods.
Changes from baseline in concentration of blood and fecal Metabolomics | 0 and 14 weeks
  Concentration of blood and fecal metabolomics will be measured using reverse phase liquid chromatography quadrupole time of flight tandem mass spectroscopy (RPLC-QTOF-MS/MS)

CONTACTS AND LOCATIONS:
Overall Officials: Nalini Kaul, PhD, Principal Investigator — Source Nutraceutical, Inc.
Locations (1):
- Hill Top Research, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No